CLINICAL TRIAL: NCT06907719
Title: Strong Fathers, Stronger Families Program Evaluation
Brief Title: Strong Fathers, Stronger Families Healthy Marriage and Responsible Fatherhood Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Seedco: Strong Fathers, Stronger Families (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: #2021/03/41
Record Dates: First submitted 2025-03-21; First posted 2025-04-02 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Fathers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Services (Experimental): Primary Services Participants receive 40 hours of the Blueprint and 24/7 Dad curricula over the course of ten weeks.
  Interventions: Other: Primary Services

INTERVENTIONS:
Other: Primary Services — Participants receive 40 hours of the Blueprint and 24/7 Dad curricula over the course of ten weeks.

SUMMARY:
The purpose of this descriptive study is to explore whether there is an association between participation in the Strong Fathers, Stronger Families program and improvements in outcomes related to parenting, co-parenting, and economic stability. Participants are surveyed at program entry and program exit, and changes in participant attitudes are assessed over time.

DETAILED DESCRIPTION:
This study is a descriptive evaluation of the Strong Fathers, Stronger Families program offered to fathers in the Memphis metropolitan area. Program participants are informed about the study and asked to provide consent to participate in the evaluation of the ten-week program. Consenting participants complete surveys at program enrollment and program exit, and survey data is used to determine if program participation is associated with short-term changes in attitudes and behaviors among participants. Changes in parenting, co-parenting, and economic stability outcomes are assessed by comparing survey answers before and after participating in 40 hours of the Blueprint and 24/7 Dad curricula.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and older)
* With children ages 0-24
* Father/father figure
* Reside in Memphis metropolitan area

Exclusion Criteria:

* Minor (under the age of 18)
* Not a father/father figure
* Children older than 24 years old
* Reside outside of Memphis metropolitan area

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 996 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation and Research
Locations (1):
- Seedco-Midsouth, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Services
Started | 996
Completed | 996
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary Services
Number analyzed (Participants) | 996
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 979
  >=65 years | 17
Age, Continuous [Mean (Full Range); unit: years] | 37.45 [18 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 936
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 797
  White | 179
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: 1) Healthy Parenting Behaviors Measurement #1
Description: Will participants report significantly healthier parenting behavior at program exit, as compared to responses at baseline?
  Items measured include:
  Parenting behavior measured with:
  13 items depending on child age - frequency of key behaviors with participant's youngest child (categorical, 5-point scale)
  Measured on the parenting behavior scale #1 as:
  1 = never, 2 = 1 to 2 days per month, 3 = 3 or 4 days per month, 4 = 2 or 3 days per week, 5 = every day or almost every day
  The higher the rating, the better the score.
  The construct is created by adding all scores together and dividing by 13. The higher the score on a scale of 1-5, the better the outcome. The lower the score, the worse the outcome.
  maximum score: 5.0, minimum score: 1.0
Time Frame: change from baseline in parenting behaviors (interactions with child) from enrollment to program exit (10 weeks).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 342
score on scale
  mean at baseline | 3.92 (.945)
  mean at follow-up | 3.97 (.883)

2. Primary Outcome: 2) Healthy Co-parenting Behaviors Measurement #1
Description: Will participants report significantly healthier co-parenting behavior at program exit, as compared to responses at baseline?
  Items measured include:
  5 items: frequency of agreement with key co-parenting behaviors (categorical, 5-point scale)
  Measured on the co-parenting behavior scale #1 as:
  1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree
  The construct is created by adding all scores together and dividing by 11. The higher the score on a scale of 1-5, the better the outcome. The lower the score, the worse the outcome.
  maximum score: 5.0, minimum score: 1.0
Time Frame: change from baseline in co-parenting behaviors (interactions with co-parent) from enrollment to program exit (10 weeks).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 469
score on scale
  mean at baseline | 3.61 (1.26)
  mean at follow-up | 3.70 (1.20)

3. Primary Outcome: 3) Economic Stability Measurement #1
Description: Will participants report significantly healthier economic stability at program exit, as compared to responses at baseline?
  Items measured include:
  1 items: yes or no questions for have checking/savings account (dichotomous)
  1=yes, 0=no
Time Frame: change from baseline in economic stability from enrollment to program exit (10 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Services
Number analyzed (Participants) | 711
Participants
  have checking account at baseline | 98
  have checking account at follow-up | 380

4. Primary Outcome: 4) Economic Stability Measurement #2
Description: Will participants report significantly healthier economic stability at program exit, as compared to responses at baseline?
  Items measured include:
  1 item: frequency of difficulty paying bills (categorical, 4-point scale)
  Measured on the economic stability scale #1 as:
  1 = never, 2 = once in a while, 3 = somewhat often, 4 = very often The lower the score, the better the outcome.
Time Frame: change from baseline in economic stability from enrollment to program exit (10 weeks).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 718
score on scale
  mean at baseline | 2.64 (1.005)
  mean at follow-up | 2.87 (.931)

ADVERSE EVENTS:
Time Frame: length of study involvement: 10 weeks
Description: The definitions of adverse events do not differ from the clinicaltrials.gov definitions.
Arm/Group | Primary Services
All-Cause Mortality (participants affected / at risk) | 0/996
Serious Adverse Events (participants affected / at risk) | 0/996
Other Adverse Events (participants affected / at risk) | 0/996

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT06907719/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT06907719/SAP_001.pdf